CLINICAL TRIAL: NCT05187364
Title: BioWare to Enhance Treatment for Alcohol Use Disorder and Posttraumatic Stress Disorder
Brief Title: BioWare for AUD and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Amber Jarnecke, Research Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00115253
Record Dates: First submitted 2021-12-28; First posted 2022-01-11 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: PTSD; Alcohol Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPE Therapy Arm (Experimental): Concurrent Treatment of PTSD and Substance Use Disorders using Prolonged Exposure (COPE)
  Interventions: Behavioral: COPE

INTERVENTIONS:
Behavioral: COPE — The COPE therapy is a talk-therapy in which individuals are asked about their trauma, alcohol use, mood, and behavior. The therapy occurs over 12 sessions and will be paired with a telehealth technology system to determine if it enhances the COPE therapy. The telehealth system is worn on the arm and hand during the out-of-office COPE homework assignments. It consists of a small camera (about the size of a pencil eraser), Bluetooth earpiece with microphone, monitors to measure and record heart rate and skin conductance, and a breathalyzer to assess blood alcohol content. The device will connect to an application on password protected cell phone that will monitor and record the above listed information as well as reported subjective units of distress and craving. A study coach will virtually guide participants through one out-of-office assignment per week using this technology. Interviews and surveys will be collected at study baseline and weekly during treatment.

SUMMARY:
This study examines the ability of an innovative telehealth technology system to enhance Concurrent Treatment of PTSD and Substance Use Disorders using Prolonged Exposure (COPE) talk-therapy for individuals with posttraumatic stress disorder (PTSD) and alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; aged 18-70 years.
2. Able to provide written informed consent.
3. Meet DSM-5 diagnostic criteria for current moderate to severe alcohol use disorder.
4. Meet DSM-5 diagnostic criteria for current PTSD.
5. Participants taking psychotropic medications will be required to be maintained on a stable dose for at least 4 weeks before study initiation.

Exclusion Criteria:

1. Meet DSM-5 criteria for a history of or current psychotic or bipolar disorders.
2. Current suicidal or homicidal ideation and intent.
3. Psychotropic medications which have been initiated during the past 4 weeks.
4. Acute alcohol withdrawal.
5. Pregnancy or breastfeeding for people of childbearing potential.
6. Currently enrolled in evidence based behavioral treatment for AUD or PTSD.
7. Implanted electronic devices of any kind, including pacemakers, electronic infusion pumps, stimulators, defibrillators or similar.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber M Jarnecke, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COPE Therapy Arm
Started | 4
Completed | 1
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | COPE Therapy Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.00 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Clinician-Administered PTSD Scale for DSM-5 [Mean (Standard Deviation); unit: units on a scale] — The Clinician-Administered PTSD Scale for DSM-5 is a structured interview assessment of PTSD symptoms over the past month.
  Scale ranges from 0-80, such that higher scores are indicative of greater PTSD symptom severity.
  units on a scale | 36.50 (4.51)
PTSD Checklist for DSM-5 [Mean (Standard Deviation); unit: units on a scale] — PTSD Checklist for DSM-5 is a self-report measure of PTSD symptoms over the past week.
  Scale ranges from 0-80, such that higher scores are indicative of greater PTSD symptom severity. This scale has a suggested cutoff score of 31-33 for a provisional diagnosis of PTSD. Population: One participant did not complete this measure at baseline
  units on a scale
    number analyzed (Participants) | 3
    (all) | 50.00 (5.57)
Percent Days Drinking (Timeline Followback) [Mean (Standard Deviation); unit: percent of days] — Percent days drinking was assessed via a 60-day Timeline Followback assessment. Higher values are indicative of a greater percentage of drinking days in the 60 prior to the assessment.
  percent of days | 41.23 (35.73)
Alcohol Use Disorder Identification Test [Mean (Standard Deviation); unit: units on a scale] — The Alcohol Use Disorder Identification Test is a self-report measure of alcohol use problems over past year.
  Scale ranges from 0-40, such that higher scores are indicative of more alcohol use problems. Scores in the 0-7 indicate low-risk consumption, scores in the 8-14 range indicate hazardous or harmful alcohol consumption, and scores at 15 or greater indicate likelihood of moderate-to-severe alcohol use disorder. Population: One participant did not complete this measure at baseline
  units on a scale
    number analyzed (Participants) | 3
    (all) | 27.67 (12.01)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Turn on and Off Equipment in 5 Minutes or Less
Description: Feasibility is 80% of participants turning on and off equipment in 5 minutes or less
Time Frame: In-Session Visit (approximately 1 week from baseline)
Population: Two enrolled participant completed this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | COPE Therapy Arm
Number analyzed (Participants) | 2
Participants | 2

2. Primary Outcome: System Usability Scale
Description: The System Usability Scale measures how usable and acceptable a product is. This scale ranges from 0-100 with higher scores being indicative of greater usability/acceptability. A mean score of 68 or greater is considered acceptable.
Time Frame: Week 12
Population: Two enrolled participants completed this assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COPE Therapy Arm
Number analyzed (Participants) | 2
units on a scale | 90.00 (7.07)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant over the course of their COPE therapy treatment (i.e., up to 12 session that could take place over 6 months).
Arm/Group | COPE Therapy Arm
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COPE Therapy Arm (N=4)
Common Cold (Infections and infestations) | 1 (1) — Common cold symptoms - found unrelated to intervention and study procedures
Stomach bug (Infections and infestations) | 1 (1) — Stomach bug symptoms - found unrelated to intervention and study procedures
COVID-19 (Infections and infestations) | 1 (1) — COVID-19 infection - found unrelated to intervention and study procedures

LIMITATIONS AND CAVEATS:
Limitations from this pilot trial include the small sample size, that some participants dropped out from the study without completing the full course of study treatment, and that not all participants were able (either due to study dropout or due to technological equipment failure) to complete all primary outcome assessments. As such, results should be interpreted with these limitations in mind.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT05187364/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT05187364/ICF_001.pdf